CLINICAL TRIAL: NCT01150123
Title: A Phase Ib Randomized, Observer-Blind, Controlled, Single Center, Dose-Ranging Study of a Group B Streptococcus Vaccine in Healthy Women 18-40 Years of Age
Brief Title: Safety and Immunogenicity of a Group B Streptococcus Vaccine in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V98_06
Record Dates: First submitted 2010-03-31; First posted 2010-06-24 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Group B Streptococcus
Keywords: Group B streptococcus; GBS; Vaccine; Group B streptococcus (GBS) disease
MeSH Terms: conditions — Guillain-Barre Syndrome; Disease | interventions — Vaccines

STUDY DESIGN:
Who Masked: Investigator

ARMS (9):
- 5 µg_No Adj (Experimental): Subjects received either 1 or 2 doses of active vaccine (5 µg) without any adjuvant
  Interventions: Biological: Group B streptococcus (GBS) vaccine- low dose
- 20 µg_No Adj (Experimental): Subjects received either 1 or 2 doses of active vaccine (20 µg) without any adjuvant.
  Interventions: Biological: Group B streptococcus (GBS) vaccine- High dose
- 5 µg_Alum (Experimental): Subjects received either 1 or 2 doses of active vaccine (5 µg) with Alum adjuvant.
  Interventions: Biological: Group B streptococcus (GBS) vaccine- low dose
- 20 µg_Alum (Experimental): Subjects received either 1 or 2 doses of active vaccine (5 µg) with Alum adjuvant.
  Interventions: Biological: Group B streptococcus (GBS) vaccine- High dose
- 5 µg_MF59-H (Experimental): Subjects received either 1 or 2 doses of active vaccine (5 µg) adjuvanted with 4.87 mg of MF59
  Interventions: Biological: Group B streptococcus (GBS) vaccine- low dose
- 20 µg_MF59-H (Experimental): Subjects received either 1 or 2 doses of active vaccine (20 µg) adjuvanted with 4.87 mg of MF59
  Interventions: Biological: Group B streptococcus (GBS) vaccine- High dose
- 5 µg_MF59-F (Experimental): Subjects received either 1 or 2 doses of active vaccine (5 µg) adjuvanted with 9.75 mg of MF59
  Interventions: Biological: Group B streptococcus (GBS) vaccine- low dose
- 20 µg_MF59-F (Experimental): Subjects received either 1 or 2 doses of active vaccine (20 µg) adjuvanted with 9.75 mg of MF59
  Interventions: Biological: Group B streptococcus (GBS) vaccine- High dose
- Placebo (Placebo Comparator): Subjects received 2 injections of placebo administered 1 month apart
  Interventions: Biological: Placebo- Saline

INTERVENTIONS:
Biological: Group B streptococcus (GBS) vaccine- low dose
  Arms: 5 µg_Alum; 5 µg_MF59-F; 5 µg_MF59-H; 5 µg_No Adj
Biological: Group B streptococcus (GBS) vaccine- High dose
  Arms: 20 µg_Alum; 20 µg_MF59-F; 20 µg_MF59-H; 20 µg_No Adj
Biological: Placebo- Saline
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and immunogenicity of a Group B Streptococcus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females 18-40 years of age inclusive.

Exclusion Criteria:

* Individuals who are pregnant or nursing.
* Individuals who have had a previous immunization with a vaccine containing streptococcus antigens or any vaccine within 30 days of enrollment through 30 days of study completion.
* Individuals with a history of severe allergic reactions after previous vaccination
* Individuals with designated blood tests that are not within normal range

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 678 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis
Locations (1):
- Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels G, Maes C, Willekens J, De Boever F, de Rooij R, Martell L, Bedell L, Wittke F, Slobod K, Dull P. A randomized, observer-blind Phase Ib study to identify formulations and vaccine schedules of a trivalent Group B Streptococcus vaccine for use in non-pregnant and pregnant women. Vaccine. 2016 Apr 4;34(15):1786-91. doi: 10.1016/j.vaccine.2016.02.044. Epub 2016 Mar 5. PMID 26928074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one center in Belgium
Pre-assignment Details: Group1: 5 µg-1Inj-No Adj, 5 µg-2Inj-No Adj, 20 µg-1Inj-No Adj, 20 µg-2Inj-No Adj (Cohort 1), 5 µg-1Inj-Alum, 5 µg-2Inj-Alum, 20 µg-1Inj-Alum, 20 µg-2Inj-Alum (Cohort 2).
  Group 2: 5 µg-1Inj-MF59_F, 5 µg-2Inj-MF59_F, 20 µg-1Inj-MF59_F, 20 µg-2Inj-MF59_F (Cohort 3), 5 µg-1Inj-MF59_H, 5 µg-2Inj-MF59_H, 20 µg-1Inj-MF59_H, 20 µg-2Inj-MF59_H (Cohort 4)
Groups:
- 5 µg-1 Inj - No Adj: Subjects received single active vaccine injection (5 µg) without any adjuvant followed by a placebo administered 1 month apart
- 5 µg-2 Inj - No Adj: Subjects received two identical active vaccine injections (5 µg) without any adjuvant administered 1 month apart
- 20 µg-1 Inj - No Adj: Subjects received single active vaccine injection (20 µg) without any adjuvant followed by a placebo administered 1 month apart
- 20 µg-2 Inj - No Adj: Subjects received two identical active vaccine injections (20 µg) without any adjuvant administered 1 month apart
- 5 µg-1 Inj - Alum: Subjects received single active vaccine injection (5 µg) with adjuvant followed by a placebo administered 1 month apart
- 5 µg-2 Inj - Alum: Subjects received two identical active vaccine injections (5 µg) with adjuvant administered 1 month apart
- 20 µg-1 Inj - Alum: Subjects received single active vaccine injection (20 µg) with adjuvant followed by a placebo administered 1 month apart
- 20 µg-2 Inj- Alum: Subjects received two identical active vaccine injections (20 µg) with adjuvant administered 1 month apart
- Placebo - Group 1; Placebo - Group 2: Subjects received two injections of placebo administered 1 month apart
- 5 µg-1 Inj - MF59_H: Subjects received single active vaccine injection (5 µg) adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
- 5 µg-2 Inj - MF59_H: Subjects received two identical active vaccine injections (5 µg) of adjuvanted with 4.87 mg of MF59 administered 1 month apart
- 20 µg-1 Inj - MF59_H: Subjects received single active vaccine injection (20 µg) adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
- 20 µg-2 Inj - MF59_H: Subjects received two identical active vaccine injections (20 µg) adjuvanted with 4.87 mg of MF59 administered 1 month apart
- 5 µg-1 Inj - MF59_F: Subjects received single active vaccine injection (5 µg) of adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
- 5 µg-2 Inj - MF59_F: Subjects received two identical active vaccine injections (5 µg) adjuvanted with 9.75 mg of MF59 administered 1 month apart
- 20 µg-1 Inj - MF59_F: Subjects received single active vaccine injection (20 µg) adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
- 20 µg-2 Inj- MF59_F: Subjects received two identical active vaccine injections (20 µg) adjuvanted with 9.75 mg of MF59 administered 1 month apart
Period: Overall Study
Arm/Group | 5 µg-1 Inj - No Adj | 5 µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5 µg-1 Inj - Alum | 5 µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1 | 5 µg-1 Inj - MF59_H | 5 µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5 µg-1 Inj - MF59_F | 5 µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Started | 40 | 40 | 39 | 40 | 40 | 40 | 39 | 40 | 20 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 20
Completed | 37 | 38 | 35 | 37 | 37 | 34 | 39 | 37 | 15 | 39 | 38 | 39 | 37 | 40 | 40 | 39 | 40 | 19
Not Completed | 3 | 2 | 4 | 3 | 3 | 6 | 0 | 3 | 5 | 1 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2 | 2 | 5 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5μg-1 Inj - No Adj: Subjects received single active vaccine injection (5 µg) without any adjuvant followed by a placebo administered 1 month apart
- 5μg-2 Inj - No Adj: Subjects received two identical active vaccine injections (5 µg) without any adjuvant administered 1 month apart
- 20 μg-1 Inj - No Adj: Subjects received single active vaccine injection (20 µg) without any adjuvant followed by a placebo administered 1 month apart
- 20 μg-2 Inj - No Adj: Subjects received two identical active vaccine injections (20 µg) without any adjuvant administered 1 month apart
- 5μg-1 Inj - Alum: Subjects received single active vaccine injection (5 µg) with adjuvant followed by a placebo administered 1 month apart
- 5μg-2 Inj - Alum: Subjects received two identical active vaccine injections (5 µg) with adjuvant administered 1 month apart
- 20 μg-1 Inj - Alum: Subjects received single active vaccine injection (20 µg) with adjuvant followed by a placebo administered 1 month apart
- 20 μg-2 Inj- Alum: Subjects received two identical active vaccine injections (20 µg) with adjuvant administered 1 month apart
- Placebo - Group 1: Subjects received two injections of placebo administered 1 month apart t
- 5μg-1 Inj -MF59_H: Subjects received single active vaccine injection (5 µg) adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
- 5μg-2 Inj -MF59_H: Subjects received two identical active vaccine injections (5 µg) of adjuvanted with 4.87 mg of MF59 administered 1 month apart
- 20 μg-1 Inj -MF59_H: Subjects received single active vaccine injection (20 µg) adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
- 20 μg-2 Inj -MF59_H: Subjects received two identical active vaccine injections (20 µg) adjuvanted with 4.87 mg of MF59 administered 1 month apart
- 5μg-1 Inj -MF59_F: Subjects received single active vaccine injection (5 µg) of adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
- 5μg-2 Inj -MF59_F: Subjects received two identical active vaccine injections (5 µg) adjuvanted with 9.75 mg of MF59 administered 1 month apart
- 20 μg-1 Inj -MF59_F: Subjects received single active vaccine injection (20 µg) adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
- 20 μg-2 Inj-MF59_F: Subjects received two identical active vaccine injections (20 µg) adjuvanted with 9.75 mg of MF59 administered 1 month apart
- Total: Total of all reporting groups
Arm/Group | 5μg-1 Inj - No Adj | 5μg-2 Inj - No Adj | 20 μg-1 Inj - No Adj | 20 μg-2 Inj - No Adj | 5μg-1 Inj - Alum | 5μg-2 Inj - Alum | 20 μg-1 Inj - Alum | 20 μg-2 Inj- Alum | Placebo - Group 1 | 5μg-1 Inj -MF59_H | 5μg-2 Inj -MF59_H | 20 μg-1 Inj -MF59_H | 20 μg-2 Inj -MF59_H | 5μg-1 Inj -MF59_F | 5μg-2 Inj -MF59_F | 20 μg-1 Inj -MF59_F | 20 μg-2 Inj-MF59_F | Placebo - Group 2 | Total
Number analyzed (Participants) | 40 | 40 | 39 | 40 | 40 | 40 | 39 | 40 | 20 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 20 | 678
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (5.5) | 26.2 (7.2) | 25.5 (5.0) | 24.1 (4.6) | 26.5 (6.2) | 25.1 (5.3) | 25.1 (6.3) | 24.3 (6.0) | 23.5 (3.2) | 23.4 (4.1) | 23.5 (5.7) | 23.5 (5.2) | 24.7 (6.1) | 23.6 (5.0) | 24.9 (5.9) | 22.7 (4.0) | 22.9 (5.8) | 23.5 (5.3) | 24.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 39 | 40 | 40 | 40 | 39 | 40 | 20 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 20 | 678
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Specific Thresholds of Antibody Concentrations for Subjects in Enrollment Group 1
Description: The percentage of subjects achieving a specific threshold of antibody concentrations of ≥ 0.5 µg/mL as determined by ELISA at day 61 across cohorts 1 and 2 for potential use in pregnant women.
Time Frame: Day 1 and Day 61
Population: Analysis was done on primary Per Protocol Set (PPS) - The subjects who received the vaccine correctly; provided evaluable serum samples at baseline and Day 61; and had no major protocol violations as defined prior to analysis.
Measure: Number; unit: percentage of subjects
Groups:
- 5µg-1 Inj - No Adj: Subjects received single active vaccine injection (5 µg) without any adjuvant followed by a placebo administered 1 month apart
- 5µg-2 Inj - No Adj: Subjects received two identical active vaccine injections (5 µg) without any adjuvant administered 1 month apart
- 5µg-1 Inj - Alum: Subjects received single active vaccine injection (5 µg) with adjuvant followed by a placebo administered 1 month apart
- 5µg-2 Inj - Alum: Subjects received two identical active vaccine injections (5 µg) with adjuvant administered 1 month apart
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 40 | 38 | 35 | 38 | 37 | 37 | 38 | 38 | 17
percentage of subjects
  Day 1 (Serogroup Ia;N=40,33,33,35,33,32,34,35,17) | 38 | 30 | 30 | 29 | 30 | 38 | 35 | 20 | 18
  Day 61 (Serogroup Ia) | 98 | 97 | 91 | 95 | 97 | 95 | 87 | 84 | 18
  Day 1 (Serogroup Ib; N=37,33,34,35,34,32,34,32,17) | 24 | 12 | 18 | 17 | 26 | 16 | 24 | 9 | 18
  Day 61 (Serogroup Ib;N=39,38,35,38,37,37,38,36,16) | 82 | 95 | 83 | 84 | 78 | 86 | 84 | 64 | 19
  Day 1 (Serogroup III;N=40,38,35,38,37,36,38,38,17) | 18 | 13 | 11 | 13 | 16 | 28 | 16 | 18 | 12
  Day 61 (SerogroupIII;N=40,37,35,38,36,37,37,37,17) | 70 | 81 | 77 | 79 | 67 | 86 | 70 | 76 | 12

2. Primary Outcome: Geometric Mean Concentrations of Serum Anti-GBS IgG Antibody Levels by Serotype at Day 61
Description: Serotype-specific (Ia, Ib & III) group B streptococcus (GBS) IgG antibody levels in healthy subjects for potential use in pregnant woman was assessed in terms of Geometric Mean Concentrations (GMCs) at Day 61 in cohorts 1 and 2.
Time Frame: Day 1 and Day 61
Population: Analysis was done on Primary PPS
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 40 | 38 | 35 | 38 | 37 | 37 | 38 | 38 | 17
µg/mL
  Day 1 (Serotype Ia; N=40,33,33,35,33,32,34,35,17) | 0.62 [0.36 to 1.08] | 0.51 [0.28 to 0.94] | 0.38 [0.21 to 0.71] | 0.45 [0.25 to 0.81] | 0.48 [0.26 to 0.87] | 0.57 [0.31 to 1.06] | 0.54 [0.29 to 0.98] | 0.37 [0.2 to 0.67] | 0.25 [0.11 to 0.59]
  Day 61 (Serotype Ia; N=40,38,35,38,37,37,38,37,17) | 20 [9.42 to 41] | 11 [5.41 to 24] | 15 [7.08 to 34] | 18 [8.34 to 37] | 14 [6.54 to 30] | 9.99 [4.67 to 21] | 9.64 [4.55 to 20] | 6.49 [3.03 to 14] | 0.25 [0.083 to 0.78]
  Day 1 (Serotype Ib; N=37,33,34,35,34,32,34,32,17 ) | 0.15 [0.089 to 0.25] | 0.11 [0.065 to 0.19] | 0.11 [0.064 to 0.19] | 0.11 [0.062 to 0.18] | 0.15 [0.088 to 0.26] | 0.12 [0.068 to 0.21] | 0.12 [0.072 to 0.21] | 0.081 [0.046 to 0.14] | 0.16 [0.072 to 0.34]
  Day 61(Serotype Ib;N=39,38,35,38,37,37,38,36,16) | 6.75 [3.21 to 14] | 4.56 [2.15 to 9.69] | 4.26 [1.95 to 9.34] | 4.45 [2.09 to 9.44] | 4.72 [2.2 to 10] | 3.85 [1.79 to 8.24] | 3.92 [1.85 to 8.32] | 2.06 [0.95 to 4.46] | 0.24 [0.075 to 0.76]
  Day 1 (Serotype III; N=40,38,35,38,37,36,38,38,17) | 0.13 [0.08 to 0.2] | 0.089 [0.056 to 0.14] | 0.087 [0.054 to 0.14] | 0.077 [0.049 to 0.12] | 0.099 [0.062 to 0.16] | 0.15 [0.096 to 0.25] | 0.09 [0.057 to 0.14] | 0.12 [0.074 to 0.19] | 0.1 [0.05 to 0.2]
  Day 61(Serotype III; N=40,37,35,38,36,37,37,37,17) | 3.27 [1.6 to 6.68] | 3.23 [1.54 to 6.78] | 2.31 [1.08 to 4.95] | 2.35 [1.13 to 4.89] | 1.49 [0.7 to 3.15] | 4.3 [2.05 to 9.04] | 1.4 [0.67 to 2.94] | 3.28 [1.56 to 6.89] | 0.1 [0.035 to 0.31]

3. Secondary Outcome: Number of Participants Reporting Solicited Adverse Events (AEs) After Receiving the GBS Trivalent Vaccine in Enrollment Group 1
Description: Safety was assessed in terms of number of participants reporting solicited local and systemic adverse events after receiving trivalent GBS vaccine from day 1 to day 7 for subjects across cohorts 1 and 2.
Time Frame: Day 1 to Day 7
Population: Analysis was done on Solicited Safety Set - All subjects in the Exposed Set who provided data on post vaccination local or systemic AEs or other signs of reactogenicity.
Measure: Number; unit: participants
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 40 | 40 | 39 | 40 | 40 | 40 | 39 | 39 | 19
participants
  Any Local | 30 | 32 | 31 | 35 | 39 | 37 | 38 | 39 | 8
  Inj site Induration | 9 | 13 | 6 | 9 | 12 | 16 | 16 | 15 | 3
  Inj site swelling | 5 | 5 | 5 | 5 | 7 | 8 | 16 | 8 | 2
  Ecchymosis | 5 | 3 | 7 | 2 | 5 | 4 | 0 | 2 | 0
  Redness | 8 | 8 | 9 | 8 | 9 | 12 | 15 | 14 | 3
  Warmth | 10 | 11 | 9 | 13 | 11 | 14 | 11 | 16 | 1
  Inj site Pain | 28 | 28 | 31 | 34 | 39 | 37 | 38 | 39 | 7
  Any Systemic | 25 | 21 | 22 | 28 | 27 | 20 | 29 | 21 | 11
  Chills | 3 | 2 | 5 | 2 | 3 | 1 | 4 | 4 | 3
  Nausea | 6 | 5 | 8 | 5 | 7 | 6 | 5 | 4 | 1
  Malaise | 7 | 6 | 11 | 11 | 7 | 9 | 12 | 9 | 2
  Myalgia | 6 | 1 | 7 | 8 | 3 | 5 | 8 | 6 | 2
  Arthralgia | 2 | 1 | 3 | 2 | 3 | 3 | 3 | 6 | 0
  Headache | 16 | 15 | 13 | 18 | 19 | 17 | 19 | 11 | 7
  Fatigue | 18 | 9 | 18 | 21 | 19 | 13 | 17 | 13 | 6
  Rash | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Fever (≥ 38C) | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 0

4. Primary Outcome: Geometric Mean Ratios of Serum Group B Streptococcus IgG Antibody Levels By Serotype
Description: Geometric mean ratios (GMRs) relative to baseline (Day 1) of serotype-specific (Ia, Ib, III) GBS IgG antibody levels measured at Day 61 for subjects across cohorts 1 and 2.
Time Frame: Day 61/Day 1
Population: Analysis was done on Primary PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | 5 µg-1 Inj - No Adj | 5 µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5 µg-1 Inj - Alum | 5 µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 40 | 37 | 34 | 38 | 36 | 36 | 37 | 37 | 17
Ratios
  serotype Ia; N=40,33,32,35,33,32,34,35,17 | 32 [19 to 53] | 28 [16 to 50] | 37 [21 to 66] | 45 [26 to 78] | 36 [20 to 64] | 23 [13 to 42] | 25 [14 to 44] | 19 [11 to 33] | 1.01 [0.46 to 2.24]
  Serotype Ib; N=37,33,33,35,34,32,34,31,16 | 47 [29 to 77] | 46 [27 to 78] | 39 [23 to 66] | 47 [28 to 79] | 38 [22 to 63] | 32 [19 to 54] | 33 [20 to 55] | 23 [13 to 39] | 1.55 [0.73 to 3.28]
  Serotype III | 26 [16 to 43] | 36 [22 to 61] | 26 [15 to 45] | 30 [18 to 50] | 15 [8.71 to 25] | 30 [18 to 50] | 16 [9.48 to 26] | 30 [18 to 50] | 1.13 [0.52 to 2.46]

5. Primary Outcome: Percentage of Subjects Achieving Specific Thresholds of Antibody Concentrations for Subjects in Enrollment Groups 1 & 2
Description: The percentage of subjects achieving a specific threshold of antibody concentrations of ≥ 0.5 µg/mL at day 361 across all the cohorts for potential use in non-pregnant women.
Time Frame: Day 1 and Day 361
Population: Analysis was done on Co-primary PPS - The subjects who received the vaccine correctly; provided evaluable serum samples at baseline and Day 361; and had no major protocol violations as defined prior to analysis
Measure: Number; unit: percentage of subjects
Groups:
- 5µg-1 Inj - MF59_H: Subjects received single active vaccine injection (5 µg) adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
- 5µg-2 Inj - MF59_H: Subjects received two identical active vaccine injections (5 µg) of adjuvanted with 4.87 mg of MF59 administered 1 month apart
- 5µg-1 Inj - MF59_F: Subjects received single active vaccine injection (5 µg) of adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
- 5µg-2 Inj - MF59_F: Subjects received two identical active vaccine injections (5 µg) adjuvanted with 9.75 mg of MF59 administered 1 month apart
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1 | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 40 | 32 | 32 | 35 | 34 | 33 | 34 | 36 | 17 | 37 | 38 | 38 | 39 | 38 | 37 | 38 | 39 | 20
percentage of subjects
  Day 1 (Serogroup Ia) | 38 | 28 | 28 | 29 | 35 | 39 | 35 | 22 | 18 | 30 | 29 | 16 | 28 | 29 | 38 | 21 | 31 | 20
  Day 361 (Serogroup Ia) | 85 | 78 | 88 | 86 | 86 | 92 | 79 | 75 | 14 | 78 | 82 | 76 | 95 | 69 | 92 | 76 | 90 | 20
  Day 1 (Serogroup Ib) | 24 | 13 | 15 | 17 | 26 | 15 | 24 | 9 | 18 | 24 | 15 | 6 | 26 | 23 | 19 | 6 | 11 | 24
  Day 361 (Serogroup Ib) | 95 | 92 | 91 | 97 | 92 | 100 | 100 | 89 | 46 | 92 | 100 | 87 | 97 | 95 | 97 | 100 | 100 | 22
  Day 1 (Serogroup III) | 18 | 14 | 12 | 13 | 16 | 30 | 16 | 18 | 12 | 14 | 11 | 5 | 8 | 14 | 14 | 11 | 8 | 0
  Day 361 (Serogroup III) | 85 | 84 | 82 | 95 | 76 | 95 | 87 | 89 | 20 | 86 | 95 | 92 | 100 | 87 | 100 | 89 | 92 | 6

6. Primary Outcome: Geometric Mean Concentrations of Serum Anti-GBS IgG Antibody Levels by Serotype at Day 361
Description: Serotype-specific (Ia, Ib & III) GBS IgG antibody levels in healthy subjects for potential use in non-pregnant woman was assessed in terms of GMCs at Day 361 across all cohorts.
Time Frame: Day 1 and Day 361
Population: Analysis was done on Co-Primary PPS
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 5 µg-1 Inj - No Adj | 5 µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5 µg-1 Inj - Alum | 5 µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1 | 5 µg-1 Inj - MF59_H | 5 µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5 µg-1 Inj - MF59_F | 5 µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 40 | 37 | 34 | 38 | 38 | 37 | 38 | 39 | 17 | 37 | 38 | 38 | 39 | 39 | 37 | 38 | 39 | 20
µg/mL
  Day1(Serotype Ia) | 0.62 [0.36 to 1.07] | 0.45 [0.25 to 0.84] | 0.36 [0.2 to 0.67] | 0.45 [0.25 to 0.8] | 0.53 [0.29 to 0.96] | 0.62 [0.34 to 1.14] | 0.54 [0.3 to 0.97] | 0.37 [0.21 to 0.66] | 0.25 [0.11 to 0.58] | 0.54 [0.32 to 0.91] | 0.43 [0.25 to 0.72] | 0.27 [0.16 to 0.45] | 0.36 [0.22 to 0.61] | 0.44 [0.26 to 0.73] | 0.46 [0.27 to 0.79] | 0.36 [0.21 to 0.6] | 0.45 [0.27 to 0.75] | 0.34 [0.17 to 0.7]
  Day361(Serotype Ia) | 5.86 [2.93 to 12] | 3.78 [1.85 to 7.72] | 4 [1.9 to 8.41] | 4.6 [2.25 to 9.38] | 5.83 [2.86 to 12] | 5.22 [2.56 to 11] | 3.78 [1.87 to 7.65] | 2.94 [1.43 to 6.05] | 0.26 [0.08 to 0.81] | 3.62 [1.84 to 7.13] | 3.04 [1.56 to 5.93] | 2.13 [1.09 to 4.15] | 7.19 [3.72 to 14] | 2.65 [1.37 to 5.12] | 7.32 [3.72 to 14] | 2.67 [1.36 to 5.24] | 4.41 [2.28 to 8.52] | 0.31 [0.12 to 0.77]
  Day1(Serotype Ib) | 0.15 [0.089 to 0.25] | 0.12 [0.066 to 0.2] | 0.099 [0.058 to 0.17] | 0.11 [0.062 to 0.18] | 0.15 [0.085 to 0.25] | 0.12 [0.069 to 0.2] | 0.12 [0.073 to 0.21] | 0.079 [0.046 to 0.14] | 0.16 [0.073 to 0.33] | 0.12 [0.071 to 0.21] | 0.1 [0.058 to 0.17] | 0.07 [0.04 to 0.12] | 0.11 [0.062 to 0.18] | 0.15 [0.083 to 0.26] | 0.11 [0.065 to 0.2] | 0.077 [0.044 to 0.13] | 0.09 [0.053 to 0.15] | 0.1 [0.048 to 0.22]
  Day361(Serotype Ib) | 4.03 [2.38 to 6.83] | 3.7 [2.15 to 6.36] | 2.86 [1.62 to 5.03] | 3.82 [2.22 to 6.58] | 3.13 [1.82 to 5.38] | 4.59 [2.67 to 7.89] | 3.38 [1.98 to 5.77] | 2.45 [1.41 to 4.24] | 0.81 [0.33 to 2.03] | 2.67 [1.53 to 4.66] | 3.81 [2.19 to 6.61] | 1.88 [1.08 to 3.27] | 5.53 [3.21 to 9.54] | 3.18 [1.85 to 5.48] | 5.19 [2.97 to 9.08] | 3.9 [2.23 to 6.82] | 3.64 [2.11 to 6.27] | 0.18 [0.079 to 0.39]
  Day1(serotype III) | 0.13 [0.08 to 0.2] | 0.091 [0.057 to 0.15] | 0.089 [0.055 to 0.15] | 0.077 [0.049 to 0.12] | 0.1 [0.064 to 0.16] | 0.16 [0.1 to 0.26] | 0.09 [0.057 to 0.14] | 0.12 [0.074 to 0.19] | 0.1 [0.05 to 0.2] | 0.1 [0.066 to 0.17] | 0.079 [0.05 to 0.13] | 0.058 [0.037 to 0.092] | 0.067 [0.042 to 0.11] | 0.1 [0.066 to 0.16] | 0.11 [0.067 to 0.17] | 0.078 [0.049 to 0.12] | 0.093 [0.059 to 0.15] | 0.068 [0.036 to 0.13]
  Day361(Serotype III) | 3.05 [1.78 to 5.2] | 2.71 [1.57 to 4.69] | 2.45 [1.38 to 4.34] | 2.78 [1.61 to 4.81] | 1.77 [1.02 to 3.07] | 4.48 [2.59 to 7.76] | 1.77 [1.03 to 3.03] | 3.46 [1.98 to 6.04] | 0.13 [0.054 to 0.3] | 2.33 [1.42 to 3.8] | 2.67 [1.64 to 4.34] | 2.06 [1.27 to 3.34] | 4.5 [2.78 to 7.26] | 2.62 [1.62 to 4.23] | 4.99 [3.05 to 8.17] | 3.07 [1.87 to 5.02] | 3.51 [2.17 to 5.67] | 0.076 [0.038 to 0.15]

7. Primary Outcome: Geometric Mean Ratios of Serum Group B Streptococcus IgG Antibody Levels By Serotype at Day 361
Description: GMRs relative to baseline (Day 1) of serotype-specific (Ia, Ib, III) GBS IgG antibody levels in healthy subjects for potential use in non-pregnant women, measured at Day 361 across all cohorts.
Time Frame: Day 1 and day 361
Population: Analysis was done on Co-Primary PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1 | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 39 | 37 | 33 | 37 | 37 | 36 | 38 | 36 | 14 | 37 | 38 | 38 | 39 | 38 | 37 | 37 | 39 | 20
Ratios
  Day361/Day1(Serotype Ia) | 9.13 [5.74 to 15] | 10 [6.09 to 17] | 9.89 [5.87 to 17] | 15 [8.9 to 24] | 14 [8.3 to 23] | 11 [6.58 to 18] | 8.93 [5.43 to 15] | 9.54 [5.8 to 16] | 0.93 [0.43 to 2.01] | 6.75 [4.44 to 10] | 7.15 [4.73 to 11] | 7.99 [5.29 to 12] | 20 [13 to 30] | 6.17 [4.09 to 9.33] | 16 [10 to 24] | 7.29 [4.8 to 11] | 9.83 [6.54 to 15] | 0.9 [0.51 to 1.59]
  Day361/Day1(Serotype Ib) | 28 [19 to 40] | 37 [26 to 55] | 26 [18 to 38] | 38 [26 to 55] | 23 [16 to 34] | 38 [26 to 55] | 27 [19 to 39] | 30 [21 to 44] | 3.97 [2.19 to 7.19] | 23 [16 to 33] | 37 [26 to 53] | 27 [18 to 39] | 54 [38 to 76] | 26 [18 to 37] | 45 [31 to 66] | 49 [34 to 71] | 35 [25 to 50] | 1.75 [1.04 to 2.94]
  Day361/Day1(Serotype III) | 24 [16 to 35] | 30 [20 to 45] | 27 [17 to 41] | 35 [23 to 53] | 17 [12 to 26] | 30 [20 to 45] | 20 [13 to 29] | 31 [20 to 47] | 1.4 [0.72 to 2.72] | 22 [15 to 33] | 35 [23 to 53] | 35 [24 to 53] | 65 [44 to 97] | 26 [18 to 40] | 45 [30 to 68] | 38 [26 to 58] | 38 [26 to 56] | 1.24 [0.7 to 2.21]

8. Secondary Outcome: Number of Participants Reporting Solicited AEs After Receiving the GBS Trivalent Vaccine in Enrollment Group 2
Description: Safety was assessed in terms of number of participants reporting solicited local and systemic adverse events after receiving GBS vaccine from day 1 to day 7 for subjects in cohorts 3 and 4.
Time Frame: Day 1 to Day 7
Population: Analysis was done on Solicited Safety Set
Measure: Number; unit: participants
Groups:
- 5µg-1 Inj - MF59_H: Subjects received single active vaccine injection adjuvanted with 4.87 mg of MF59 followed by a placebo administered 1 month apart
Arm/Group | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 20
participants
  Any Local | 33 | 37 | 36 | 40 | 37 | 38 | 39 | 39 | 8
  Inj site Induration | 5 | 12 | 7 | 12 | 8 | 9 | 14 | 14 | 3
  Inj site swelling | 2 | 9 | 7 | 11 | 8 | 10 | 7 | 13 | 2
  Ecchymosis | 2 | 4 | 4 | 2 | 5 | 4 | 5 | 5 | 2
  Redness | 3 | 11 | 8 | 8 | 6 | 8 | 7 | 17 | 4
  Warmth | 6 | 17 | 14 | 21 | 12 | 14 | 17 | 21 | 6
  Inj site Pain | 32 | 35 | 35 | 40 | 37 | 37 | 39 | 39 | 5
  Any Systemic | 23 | 28 | 23 | 31 | 28 | 31 | 30 | 34 | 13
  Chills | 2 | 5 | 7 | 9 | 7 | 7 | 5 | 16 | 5
  Nausea | 8 | 8 | 6 | 10 | 5 | 10 | 8 | 13 | 5
  Malaise | 11 | 17 | 13 | 13 | 17 | 15 | 17 | 20 | 6
  Myalgia | 6 | 11 | 8 | 10 | 14 | 10 | 7 | 17 | 2
  Arthralgia | 1 | 3 | 5 | 3 | 3 | 4 | 4 | 7 | 1
  Headache | 13 | 19 | 14 | 23 | 14 | 23 | 22 | 30 | 10
  Fatigue | 17 | 18 | 18 | 21 | 25 | 20 | 20 | 22 | 9
  Rash | 0 | 1 | 2 | 1 | 2 | 1 | 3 | 1 | 0
  Fever (≥ 38C) | 0 | 1 | 2 | 1 | 5 | 1 | 4 | 6 | 0

9. Secondary Outcome: Number of Participants Reporting Unsolicited AE After Receiving GBS Trivalent Vaccine in Enrollment Group 1
Description: Safety was assessed in terms of number of participants with unsolicited AEs after receiving GBS trivalent vaccine, reported from day 1 to day 721 across subjects in cohorts 1 and 2.
Time Frame: Day 1 through Day 721
Population: Analysis was done on unsolicited safety set - All subjects in the Exposed Set who provided information about postvaccination unsolicited AEs.
Measure: Number; unit: participants
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 40 | 40 | 39 | 40 | 40 | 40 | 39 | 39 | 19
participants
  Any AEs | 32 | 33 | 31 | 27 | 32 | 30 | 33 | 32 | 16
  At least possibly related AEs | 8 | 11 | 11 | 11 | 4 | 6 | 7 | 5 | 0
  Serious AEs | 1 | 1 | 0 | 2 | 6 | 2 | 2 | 0 | 2
  Medically attended AEs | 25 | 24 | 23 | 18 | 26 | 24 | 28 | 27 | 11

10. Secondary Outcome: Number of Participants Reporting Unsolicited AE After Receiving GBS Trivalent Vaccine in Enrollment Group 2
Description: Safety was assessed in terms of number of participants with unsolicited AEs after receiving GBS trivalent vaccine, reported from day 1 to day 721 across subjects in cohorts 3 and 4.
Time Frame: Day 1 through Day 721
Population: Analysis was done on Unsolicited Safety Set.
Measure: Number; unit: participants
Groups:
- 5µg-2 Inj - MF59_F: Subjects received single active vaccine injection (5 µg) of adjuvanted with 9.75 mg of MF59 followed by a placebo administered 1 month apart
Arm/Group | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 20
participants
  Any AEs | 30 | 34 | 36 | 38 | 29 | 35 | 34 | 32 | 16
  At least possibly related AEs | 0 | 6 | 5 | 6 | 4 | 2 | 9 | 13 | 1
  Serious AEs | 2 | 2 | 0 | 3 | 3 | 2 | 6 | 2 | 1
  Medically attended AEs | 27 | 26 | 26 | 27 | 22 | 28 | 27 | 26 | 10

11. Secondary Outcome: Persistence of Antibody Response in Terms of Geometric Mean Concentrations by Serotype for Subjects in Enrollment Group 1
Description: The persistence of Serotype-specific (Ia, Ib & III) GBS IgG antibody response was assessed by comparing ELISA responses in terms of GMCs at day 721 after the first injection for subjects enrolled in cohorts 1 and 2.
Time Frame: Day 1 and Day 721
Population: Analysis was done on secondary persistence PPS - All the subjects who provided all serum sample results from Baseline (prior to vaccination) through Day 721 within protocol required windows.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 36 | 32 | 29 | 31 | 29 | 27 | 33 | 31 | 9
µg/mL
  Day 1 (serotype Ia) | 0.63 [0.35 to 1.11] | 0.45 [0.25 to 0.83] | 0.39 [0.21 to 0.75] | 0.34 [0.19 to 0.64] | 0.55 [0.29 to 1.04] | 0.49 [0.25 to 0.95] | 0.56 [0.31 to 1.01] | 0.34 [0.18 to 0.63] | 0.37 [0.12 to 1.16]
  Day 721 (Serotype Ia) | 4.69 [2.23 to 9.89] | 3.48 [1.58 to 7.67] | 3.11 [1.36 to 7.14] | 3.18 [1.42 to 7.09] | 5.1 [2.23 to 12] | 3.01 [1.27 to 7.11] | 3.69 [1.69 to 8.03] | 2.17 [0.97 to 4.85] | 0.3 [0.068 to 1.34]
  Day 1(Serotype Ib;N=32,30,28,32,29,28,28,27,6) | 0.16 [0.089 to 0.28] | 0.11 [0.061 to 0.2] | 0.094 [0.051 to 0.17] | 0.11 [0.063 to 0.2] | 0.18 [0.1 to 0.33] | 0.13 [0.069 to 0.23] | 0.14 [0.078 to 0.27] | 0.085 [0.045 to 0.16] | 0.88 [0.23 to 3.29]
  Day 721(Serotype Ib;N=32,30,28,32,29,28,28,27,6) | 2.92 [1.51 to 5.64] | 2.81 [1.42 to 5.55] | 1.71 [0.85 to 3.46] | 2.64 [1.37 to 5.1] | 2.32 [1.16 to 4.64] | 2.96 [1.47 to 5.99] | 2.55 [1.26 to 5.15] | 1.45 [0.71 to 2.97] | 1.02 [0.22 to 4.68]
  Day 1(Serotype III;N=34,33,28,34,30,30,34,31,6) | 0.14 [0.083 to 0.23] | 0.097 [0.058 to 0.16] | 0.094 [0.053 to 0.17] | 0.079 [0.047 to 0.13] | 0.12 [0.069 to 0.21] | 0.16 [0.095 to 0.28] | 0.095 [0.057 to 0.16] | 0.12 [0.07 to 0.21] | 0.071 [0.021 to 0.24]
  Day 721(Serotype III;N=34,33,28,34,30,30,34,31,6) | 3.19 [1.77 to 5.77] | 1.89 [1.04 to 3.45] | 1.7 [0.89 to 3.27] | 2.16 [1.2 to 3.91] | 1.26 [0.67 to 2.36] | 3.87 [2.06 to 7.26] | 1.44 [0.8 to 2.6] | 2.68 [1.44 to 4.99] | 0.054 [0.013 to 0.22]

12. Secondary Outcome: Persistence of Antibody Response in Terms of Geometric Mean Concentrations by Serotype in Subjects in Enrollment Group 2
Description: The persistence of Serotype-specific (Ia, Ib & III) GBS IgG antibody response assessed by comparing ELISA responses in terms of GMCs at day 721 after the first injection for subjects enrolled in cohort 3 and 4.
Time Frame: Day 1 and Day 721
Population: Analysis was done on secondary persistence PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 35 | 34 | 34 | 34 | 36 | 33 | 37 | 36 | 18
µg/mL
  Day 1 (serotype Ia) | 0.47 [0.27 to 0.81] | 0.48 [0.27 to 0.83] | 0.28 [0.16 to 0.49] | 0.29 [0.17 to 0.51] | 0.46 [0.27 to 0.79] | 0.53 [0.3 to 0.93] | 0.37 [0.21 to 0.62] | 0.49 [0.28 to 0.84] | 0.37 [0.17 to 0.79]
  Day 721 (Serotype Ia) | 1.86 [0.9 to 3.83] | 1.97 [0.95 to 4.11] | 1.73 [0.83 to 3.6] | 3.09 [1.49 to 6.44] | 1.66 [0.82 to 3.39] | 5.06 [2.4 to 11] | 1.72 [0.85 to 3.47] | 3.32 [1.63 to 6.77] | 0.33 [0.12 to 0.9]
  Day 1(Serotype Ib;N=32,28,29,29,28,24,30,33,9) | 0.13 [0.074 to 0.23] | 0.092 [0.051 to 0.17] | 0.072 [0.04 to 0.13] | 0.1 [0.058 to 0.19] | 0.15 [0.08 to 0.27] | 0.15 [0.077 to 0.28] | 0.08 [0.045 to 0.14] | 0.094 [0.054 to 0.16] | 0.16 [0.055 to 0.46]
  Day 721(Serotype Ib;N=32,28,29,29,28,24,30,33,9) | 1.7 [0.9 to 3.22] | 1.72 [0.87 to 3.41] | 1.16 [0.59 to 2.27] | 2.99 [1.53 to 5.86] | 2.5 [1.26 to 4.96] | 4.23 [2.02 to 8.84] | 2.47 [1.28 to 4.79] | 1.93 [1.03 to 3.61] | 0.21 [0.063 to 0.7]
  Day 1(Serotype III;N=34,32,34,32,33,31,36,33,14) | 0.11 [0.068 to 0.18] | 0.082 [0.049 to 0.14] | 0.061 [0.037 to 0.1] | 0.071 [0.043 to 0.12] | 0.09 [0.054 to 0.15] | 0.12 [0.069 to 0.2] | 0.077 [0.048 to 0.12] | 0.1 [0.06 to 0.17] | 0.061 [0.028 to 0.13]
  Day721(Serotype III;N=34,32,34,32,33,31,36,33,14) | 1.72 [1 to 2.96] | 1.59 [0.91 to 2.79] | 1.29 [0.75 to 2.23] | 2.48 [1.42 to 4.33] | 2.04 [1.17 to 3.53] | 3.18 [1.8 to 5.61] | 1.78 [1.05 to 3.02] | 2.05 [1.18 to 3.56] | 0.075 [0.032 to 0.17]

13. Secondary Outcome: Geometric Mean Ratios of Serum GBS IgG Antibody Levels By Serotype for Subjects in Enrollment Group 1
Description: GMR was calculated at Day 721 relative to baseline (Day 1) of serotype-specific (Ia, Ib, III) GBS IgG antibody levels across all cohorts 1 and 2.
Time Frame: Day 1 and Day 721
Population: Analysis was done on secondary persistence PPS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1
Number analyzed (Participants) | 36 | 32 | 29 | 31 | 29 | 27 | 33 | 31 | 9
Ratios
  Day 721/Day 1(Serotype Ia) | 7.5 [4.51 to 12] | 7.67 [4.47 to 13] | 7.89 [4.48 to 14] | 9.24 [5.34 to 16] | 9.25 [5.25 to 16] | 6.15 [3.42 to 11] | 6.64 [3.9 to 11] | 6.35 [3.67 to 11] | 0.82 [0.3 to 2.26]
  Day 721/ Day 1 (Serotype Ib) | 19 [12 to 28] | 26 [17 to 40] | 18 [12 to 29] | 24 [15 to 36] | 13 [8.16 to 20] | 23 [15 to 37] | 18 [11 to 28] | 17 [11 to 27] | 1.17 [0.44 to 3.1]
  Day 721/ Day 1 (Serotype III) | 23 [15 to 35] | 19 [13 to 30] | 18 [11 to 29] | 27 [18 to 41] | 11 [6.81 to 16] | 24 [15 to 37] | 15 [10 to 23] | 22 [14 to 35] | 0.76 [0.28 to 2.06]

14. Secondary Outcome: Geometric Mean Ratios of Serum GBS IgG Antibody Levels By Serotype for Subjects in Enrollment Group 2
Description: GMR was calculated at Day 721 relative to baseline (Day 1) of serotype-specific (Ia, Ib, III) GBS IgG antibody levels across cohorts 3 and 4.
Time Frame: Day 1 and Day 721
Population: Analysis was done on secondary persistence PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Number analyzed (Participants) | 35 | 34 | 34 | 34 | 36 | 33 | 37 | 36 | 18
Ratios
  Day 721/Day 1 (Serotype Ia) | 3.98 [2.55 to 6.2] | 4.14 [2.64 to 6.5] | 6.12 [3.9 to 9.6] | 11 [6.74 to 17] | 3.61 [2.33 to 5.6] | 9.61 [6.09 to 15] | 4.7 [3.05 to 7.23] | 6.8 [4.39 to 11] | 0.89 [0.48 to 1.65]
  Day 721/Day 1 (Serotype Ib) | 13 [8.76 to 20] | 19 [12 to 29] | 16 [10 to 24] | 29 [19 to 44] | 17 [11 to 26] | 29 [18 to 45] | 31 [20 to 47] | 20 [14 to 30] | 1.31 [0.61 to 2.8]
  Day 721/Day 1 (Serotype III) | 16 [10 to 24] | 19 [12 to 30] | 21 [14 to 33] | 35 [22 to 54] | 23 [15 to 35] | 27 [17 to 43] | 23 [15 to 35] | 21 [13 to 32] | 1.22 [0.62 to 2.4]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 721
Description: All Solicited AEs are classified as systematic assessment and all unsolicited AEs are classified as non-systematic assessment.
  Safety analysis was done on As treated set.
Arm/Group | 5µg-1 Inj - No Adj | 5µg-2 Inj - No Adj | 20 µg-1 Inj - No Adj | 20 µg-2 Inj - No Adj | 5µg-1 Inj - Alum | 5µg-2 Inj - Alum | 20 µg-1 Inj - Alum | 20 µg-2 Inj- Alum | Placebo - Group 1 | 5µg-1 Inj - MF59_H | 5µg-2 Inj - MF59_H | 20 µg-1 Inj - MF59_H | 20 µg-2 Inj - MF59_H | 5µg-1 Inj - MF59_F | 5µg-2 Inj - MF59_F | 20 µg-1 Inj - MF59_F | 20 µg-2 Inj- MF59_F | Placebo - Group 2
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/40 | 0/39 | 2/40 | 6/40 | 2/40 | 2/39 | 0/40 | 2/20 | 2/40 | 2/40 | 0/40 | 3/40 | 3/40 | 2/40 | 6/40 | 2/40 | 1/20
Other Adverse Events (participants affected / at risk) | 37/40 | 38/40 | 38/39 | 39/40 | 39/40 | 39/40 | 39/39 | 39/39 | 18/19 | 38/40 | 37/40 | 40/40 | 40/40 | 39/40 | 39/40 | 40/40 | 40/40 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5µg-1 Inj - No Adj (N=40) | 5µg-2 Inj - No Adj (N=40) | 20 µg-1 Inj - No Adj (N=39) | 20 µg-2 Inj - No Adj (N=40) | 5µg-1 Inj - Alum (N=40) | 5µg-2 Inj - Alum (N=40) | 20 µg-1 Inj - Alum (N=39) | 20 µg-2 Inj- Alum (N=40) | Placebo - Group 1 (N=20) | 5µg-1 Inj - MF59_H (N=40) | 5µg-2 Inj - MF59_H (N=40) | 20 µg-1 Inj - MF59_H (N=40) | 20 µg-2 Inj - MF59_H (N=40) | 5µg-1 Inj - MF59_F (N=40) | 5µg-2 Inj - MF59_F (N=40) | 20 µg-1 Inj - MF59_F (N=40) | 20 µg-2 Inj- MF59_F (N=40) | Placebo - Group 2 (N=20)
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lyme Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eating Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniere's Disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pilonidal Cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decompression Sickness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5µg-1 Inj - No Adj (N=40) | 5µg-2 Inj - No Adj (N=40) | 20 µg-1 Inj - No Adj (N=39) | 20 µg-2 Inj - No Adj (N=40) | 5µg-1 Inj - Alum (N=40) | 5µg-2 Inj - Alum (N=40) | 20 µg-1 Inj - Alum (N=39) | 20 µg-2 Inj- Alum (N=39) | Placebo - Group 1 (N=19) | 5µg-1 Inj - MF59_H (N=40) | 5µg-2 Inj - MF59_H (N=40) | 20 µg-1 Inj - MF59_H (N=40) | 20 µg-2 Inj - MF59_H (N=40) | 5µg-1 Inj - MF59_F (N=40) | 5µg-2 Inj - MF59_F (N=40) | 20 µg-1 Inj - MF59_F (N=40) | 20 µg-2 Inj- MF59_F (N=40) | Placebo - Group 2 (N=20)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid Edema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 3 | 5 | 1 | 3 | 1 | 1 | 3 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 6 | 9 | 7 | 7 | 8 | 6 | 4 | 1 | 10 | 8 | 7 | 11 | 5 | 10 | 10 | 13 | 5
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 4 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 1
Chills (General disorders) | 3 | 2 | 5 | 2 | 3 | 1 | 4 | 4 | 3 | 2 | 5 | 7 | 9 | 7 | 7 | 5 | 16 | 5
Fatigue (General disorders) | 19 | 11 | 18 | 21 | 19 | 13 | 18 | 14 | 7 | 17 | 18 | 19 | 22 | 26 | 20 | 20 | 22 | 9
Influenza Like Illness (General disorders) | 3 | 1 | 2 | 1 | 5 | 2 | 2 | 4 | 1 | 7 | 6 | 4 | 7 | 3 | 6 | 5 | 6 | 1
Injection Site Erythema (General disorders) | 8 | 8 | 9 | 8 | 9 | 12 | 15 | 15 | 3 | 3 | 11 | 8 | 8 | 6 | 8 | 7 | 17 | 4
Injection Site Hemorrhage (General disorders) | 5 | 3 | 7 | 2 | 5 | 4 | 0 | 2 | 0 | 2 | 5 | 4 | 2 | 5 | 4 | 5 | 5 | 2
Injection Site Induration (General disorders) | 9 | 13 | 7 | 9 | 12 | 16 | 16 | 16 | 3 | 5 | 12 | 7 | 12 | 8 | 9 | 14 | 14 | 3
Injection Site Movement Impairment (General disorders) | 2 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 28 | 28 | 31 | 35 | 39 | 37 | 38 | 39 | 7 | 32 | 35 | 35 | 40 | 37 | 37 | 39 | 39 | 5
Injection Site Swelling (General disorders) | 6 | 6 | 5 | 5 | 7 | 8 | 16 | 8 | 2 | 2 | 9 | 7 | 11 | 8 | 10 | 7 | 13 | 2
Injection Site Warmth (General disorders) | 11 | 11 | 9 | 13 | 11 | 14 | 11 | 16 | 1 | 6 | 17 | 14 | 21 | 12 | 14 | 17 | 21 | 6
Malaise (General disorders) | 8 | 6 | 11 | 11 | 8 | 9 | 12 | 9 | 2 | 11 | 17 | 13 | 14 | 17 | 15 | 17 | 20 | 6
Pyrexia (General disorders) | 2 | 0 | 4 | 1 | 2 | 3 | 3 | 3 | 0 | 0 | 3 | 3 | 2 | 6 | 2 | 6 | 10 | 0
Allergy To Arthropod Bite (Immune system disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 2 | 1 | 1
Chlamydial Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coxsackie Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 3 | 0 | 4 | 0 | 3 | 1 | 2 | 1 | 2 | 3 | 2 | 1 | 3 | 2 | 0 | 2 | 2
Cytomegalovirus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 5 | 3 | 3 | 5 | 4 | 6 | 1 | 10 | 4 | 2 | 5 | 5 | 5 | 4 | 3 | 4
Oral Herpes (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 3 | 1 | 3 | 3 | 3 | 5 | 5 | 0 | 2 | 2 | 6 | 6 | 2 | 1 | 7 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 8 | 2 | 2 | 0 | 3 | 1 | 1 | 0 | 4 | 2 | 4 | 8 | 4 | 3 | 4 | 4 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 2 | 2 | 1 | 2 | 2 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 2 | 5 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 7 | 6 | 7 | 8 | 8 | 10 | 7 | 4 | 11 | 14 | 10 | 15 | 16 | 8 | 13 | 8 | 10
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 2 | 5 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 4 | 3 | 2 | 1 | 0 | 5 | 3 | 0 | 1 | 1 | 0 | 4 | 3 | 1 | 1 | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 3 | 3 | 4 | 4 | 6 | 0 | 2 | 3 | 6 | 3 | 3 | 4 | 5 | 9 | 1
Backpain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 0 | 2 | 1 | 3 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 8 | 8 | 3 | 5 | 8 | 7 | 2 | 6 | 13 | 10 | 10 | 16 | 10 | 7 | 17 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 19 | 15 | 16 | 21 | 21 | 19 | 20 | 16 | 10 | 13 | 20 | 18 | 26 | 15 | 24 | 25 | 30 | 10
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burnout Syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 4 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 2 | 1 | 6 | 3 | 3 | 5 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 2 | 2 | 3 | 3 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days